CLINICAL TRIAL: NCT02446834
Title: Research of Intensive Lifestyle Intervention for Overweight PCOS Patients With Impaired Glucose Tolerance in Their Metabolic and Reproductive Abnormalities Treatment
Brief Title: Research of Intensive Lifestyle Intervention for PCOS Patients With IGT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: [2015]018K
Record Dates: First submitted 2015-05-06; First posted 2015-05-18 (Estimated); Last update posted 2022-10-17 (Actual); Status verified 2017-11

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; intensive lifestyle intervention; IGT; drugs treatment
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Glucagon-Like Peptide-1 Receptor Agonists; Metformin; Acarbose

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (4):
- intensive lifestyle intervention (Experimental): 3 months intensive lifestyle intervention, including low GI diet and exercise.
  Interventions: Behavioral: intensive lifestyle intervention
- GLP-1 Receptor Agonists (Experimental): 3 months GLP-1 Receptor Agonists treatment
  Interventions: Drug: GLP-1 Receptor Agonists
- metformin (Experimental): 3 months metformin treatment
  Interventions: Drug: Metformin
- acarbose (Experimental): 3 months acarbose treatment
  Interventions: Drug: Acarbose

INTERVENTIONS:
Behavioral: intensive lifestyle intervention — 3 months low GI diet and exercise
  Other Names: group 1
  Arms: intensive lifestyle intervention
Drug: GLP-1 Receptor Agonists — Use GLP-1 Receptor Agonists 3 months to treat PCOS
  Other Names: group 2
  Arms: GLP-1 Receptor Agonists
Drug: Metformin — Use metformin 3 months to treat PCOS
  Other Names: group 3
  Arms: metformin
Drug: Acarbose — Use acarbose 3 months to treat PCOS
  Other Names: group 4
  Arms: acarbose

SUMMARY:
Compare the efficacy between intensive lifestyle intervention and drugs (GLP-1 Receptor Agonists, metformin and acarbose) for PCOS patients with early onset diabetes in their metabolic and reproductive abnormalities treatment; clear the treatment effect and mechanism of intensive lifestyle intervention to PCOS.

DETAILED DESCRIPTION:
We designed a non randomized control study to compare the efficacy between intensive lifestyle intervention and drugs (GLP-1 Receptor Agonists, metformin and acarbose) for PCOS patients with early onset diabetes in their metabolic and reproductive abnormalities treatment We planed to enroll 48 patients.Overweight and obese PCOS patients with newly diagnosed IGT; PCOS diagnosis based on 1990 NIH criteria. Overweight / obesity diagnostic criteria according to WHO-WPR. IGT diagnostic criteria according to 1998 WHO diagnostic criteria. Except for serious complications (cardiovascular events and recent significant kidney or lung disease within 3 months), and had high blood pressure (>160/100mmHg), blood sugar and high blood lipids (glycated hemoglobin> 11%, triglycerides >600 mg/dl).

Then we devided the 48 patients into 4 groups: intensive lifestyle intervention group, GLP-1 group, metformin group and acarbose group, and each group 12 samples. Each group use specific treatment(showed as the group name) 3 months. Before and after the intervention, the blood samples would be collected to Glucose, Insulin, GLP-1, Glucagon, sex hormones, Blood chemistry for liver and kidney function ect, as well as the image examinations.

We will compare the data of each patient, finally identify the treatment effect and mechanism of intensive lifestyle intervention to PCOS.

ELIGIBILITY:
Inclusion Criteria:

* Overweight and obese PCOS patients with newly diagnosed IGT; PCOS diagnosis based on 1990 NIH criteria. Overweight / obesity diagnostic criteria according to WHO-WPR. IGT diagnostic criteria according to 1998 WHO diagnostic criteria.

Exclusion Criteria:

* Except for serious complications (cardiovascular events and recent significant kidney or lung disease within 3 months), and had high blood pressure (>160/100mmHg), blood sugar and high blood lipids (glycated hemoglobin> 11%, triglycerides >600 mg/dl).

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
changes of Islet β-cell functions from baseline | up to 12 weeks
  Insulin and blood glucose levels

SECONDARY OUTCOMES:
Incretin | up to 12 weeks
  GLP-1, glucagon，GIP, PYY
Intra-abdominal fat distribution | up to 12 weeks
  measured by MRI
Sex Hormone | up to 12 weeks
  testosterone, estradiol, LH, and FSH

CONTACTS AND LOCATIONS:
Overall Officials: Tao Tao, MD, Study Chair — RenJi Hospital Department of Endocrinology and Metabolism
Locations (1):
- Renji Hospital Department of Endocrinology and Metabolism, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided